CLINICAL TRIAL: NCT05037929
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Astegolimab in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Astegolimab in Participants With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB43311
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — astegolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Astegolimab Q2W (Experimental): Participants will receive subcutaneous (SC) astegolimab every 2 weeks (Q2W).
  Interventions: Drug: Astegolimab
- Astegolimab Q4W (Experimental): Participants will receive alternating SC astegolimab and placebo Q2W, thus receiving astegolimab every 4 weeks (Q4W).
  Interventions: Drug: Astegolimab
- Placebo (Placebo Comparator): Participants will receive SC placebo Q2W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Astegolimab — Participants will receive SC astegolimab Q2W or Q4W.
  Arms: Astegolimab Q2W; Astegolimab Q4W
Drug: Placebo — Participants will receive SC placebo Q2W.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of astegolimab in combination with standard of care chronic obstructive pulmonary disease (COPD) maintenance therapy in patients with COPD who are former or current smokers and have a history of frequent exacerbations.

ELIGIBILITY:
Inclusion Criteria

* Documented physician diagnosis of COPD for at least 12 months
* History of frequent exacerbations, defined as having had two or more moderate or severe exacerbations occurring within a 12-month period in the 24 months prior to screening
* Post-bronchodilator FEV1 >=20 and <80% of predicted normal value at screening
* Modified Medical Research Council (dyspnea scale) (mMRC) score >=2
* Current or former smoker with a minimum of 10 pack-year history
* History of one of the following combinations of optimized, stable, standard-of-care COPD maintenance therapy for at least 4 weeks prior to screening, with no anticipated changes in therapy prior to initiation of study drug and throughout the study: Inhaled corticosteroid (ICS) plus long-acting beta-agonist (LABA); Long-acting muscarinic antagonist (LAMA) plus LABA; ICS plus LAMA plus LABA

Exclusion Criteria

* Current documented diagnosis of asthma according to the Global Initiative for Asthma guidelines or other accepted guidelines within 5 years prior to screening
* History of clinically significant pulmonary disease other than COPD
* History of long-term treatment with oxygen at >4.0 liters/minute
* Lung volume reduction surgery or procedure within 12 months prior to screening
* Participation in or planned participation in a new pulmonary rehabilitation program. Patients who are in the maintenance phase of a rehabilitation program are eligible
* History of lung transplant
* Occurrence of moderate or severe COPD exacerbation, COVID-19, upper or lower respiratory infection, pneumonia, or hospitalization of 24 hours duration within 4 weeks prior to initiation of study drug
* Treatment with oral, IV, or IM corticosteroids within 4 weeks prior to initiation of study drug
* Initiation of a methylxanthine preparation, maintenance macrolide therapy, and/or PDE4 inhibitor within 4 weeks prior to screening
* Unstable cardiac disease, myocardial infarction, or New York Heart Association Class III or IV heart failure within 12 months prior to screening

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1334 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Annualized Rate of Moderate and Severe COPD Exacerbations Over the 52-Week Treatment Period | Baseline up to Week 52

SECONDARY OUTCOMES:
Time to First Moderate or Severe COPD Exacerbation During the 52-Week Treatment Period | Baseline up to Week 52
Absolute Change from Baseline in Health-Related Quality of Life (HRQoL) at Week 52 as Assessed Through the St. George's Respiratory Questionnaire-COPD (SGRQ-C) Total Score | Baseline to Week 52
Proportion of SGRQ-C Responders at Week 52 | Baseline to Week 52
Absolute Change from Baseline in Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) (liters) at Week 52 | Baseline to Week 52
Absolute Change from Baseline in Evaluating Respiratory Symptoms in COPD (E-RS:COPD) Total Score at Week 52 | Baseline to Week 52
Annualized Rate of Severe COPD Exacerbations Over the 52-Week Treatment Period | Baseline up to Week 52
Absolute Change from Baseline in Five-Repetition Sit-to-Stand (5STS) time (seconds) at Week 52 | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (181):
- United States (34):
  - SEC Clinical Research LLC - Dothan 2 - ClinEdge - PPDS, Dothan, Alabama
  - Jasper Summit Research LLC, Jasper, Alabama
  - Pulmonary Associates of Mobile PC, Mobile, Alabama
  - Cadena Care Institute, LLC, Poway, California
  - Inst. of Healthcare Assessment, Inc., San Diego, California
  - Allianz Research Institute Inc, Westminster, California
  - National Jewish Health, Denver, Colorado
  - Clinical Site Partners - Leesburg Suite 101 - HyperCore - PPDS, Leesburg, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Clinical Site Partners - Winter Park - HyperCore - PPDS, Winter Park, Florida
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - Exordia Medical Research, Inc., Fall River, Massachusetts
  - Northern Pines Health Center PC, Buckley, Michigan
  - Revive Research Institute, Lathrup Village, Michigan
  - Cardio-Pulmonary Associates, Chesterfield, Missouri
  - Blessing Health Hannibal, Hannibal, Missouri
  - Midwest Chest Consultants, Saint Charles, Missouri
  - CARE Clinical Research, St Louis, Missouri
  - Midwest Clinical Research LLC, St Louis, Missouri
  - Sierra Clinical Research - ClinEdge - PPDS, Las Vegas, Nevada
  - American Health Research Inc., Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Carolina Research Center, Shelby, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, North Charleston, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Velocity Clinical Research Spartanburg PPDS, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - South Texas Medical Research Institute, Inc., dba TTS Research ? ClinEdge ? PPDS, Boerne, Texas
  - Baylor College of Medicine, Houston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Sherman Clinical Research - ClinEdge - PPDS, Sherman, Texas
- Argentina (17):
  - Centro Medico IPAM, Rosario, Santa Fe Province
  - Centro de Investigaciones Clínicas Belgrano, Buenos Aires
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - Fundacion Cidea, Buenos Aires
  - Centro Médico Dra de Salvo, Buenos Aires
  - CARE - Centro de Alergia y Enfermedades Respiratorias, CABA
  - Instituto de Medicina Respiratoria, IMeR, Córdoba
  - Centro de Especialidades Medicas Lobos, Lobos
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto Ave Pulmo, Mar del Plata
  - INSARES, Mendoza
  - Centro Respiratorio Quilmes, Quilmes
  - Instituto Medico Fundacion Grupo Colaborativo Rosario Investigacion y Prevencion Medica, Rosario
  - Centro Médico Respire, San Fernando
  - Instituto De Enfermedades Respiratorias E Investigacion Medica, San Juan Bautista
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Centro Integral de Medicina Respiratoria (CIMER), San Miguel de Tucumán
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - TrialsWest Pty Ltd, Spearwood, Western Australia
- Belgium (6):
  - AZ Sint-Maarten, Mechelen, Antwerpen
  - UZ Antwerpen, Edegem
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - AZ Delta, Roeselare
  - Office of Marc De Meulemeester, Thuin
  - CHU UCl Namur asbl - Site Godinne, Yvoir
- Bulgaria (12):
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases - Haskovo EOOD, Haskovo
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Dr.Nikola Penchev-Paza, Pazardzhik
  - Specialized Hospital for Active Treatment of Pulmonary Diseases- Pernik EOOD, Pernik
  - Medical center Medconsult Pleven OOD, Pleven
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Medical center Unimed EOOD, Plovdiv
  - Medical Centre Respiro OOD, Razgrad
  - Medical Center Hera EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - Medical Center New rehabilitation center EOOD, Stara Zagora
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases-Vratsa, Vratsa
- Canada (4):
  - Burlington Lung Clinic, Burlington, Ontario
  - St. Joseph's Healthcare Hamilton- Charlton Campus, Hamilton, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan
- Chile (8):
  - Centro de Investigaciones Medicas Respiratorias, Providencia, Región-MetropolitanadeSantiago
  - Centro de Investigación Curico, Curicó
  - MIRES/MYF estudios clinicos, Ñuñoa
  - Sociedad Médica SyG SpA, Providencia
  - Enroll SpA - PPDS, Providencia
  - Meditek Ltda, Santiago
  - Centro de Investigacion del Maule, Talca
  - Hospital Carlos Van Buren, Valparaíso
- Czechia (5):
  - MediTrial s.r.o., Jind?ich?v Hradec
  - Plicni Ambulance Kralupy nad Vltavou, Kralupy nad Vltavou
  - MUDr. Ilona Pavlisova s.r.o., Miroslav
  - Pneumologie Varnsdorf S.r.o., Nový Bor
  - KASMED s.r.o., Tábor
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Gentofte Hospital, Hellerup
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense
  - Sygehus Lillebælt, Vejle, Vejle
- France (3):
  - Hôpital de La Croix Rousse, Lyon
  - CHU de Nice, Nice
  - Nouvel Hôpital Civil, Strasbourg
- Germany (13):
  - Zentrum fuer Pneumologie, Onkologie und Schlafmedizin am Diako, Augsburg
  - CIMS-Studienzentrum Bamberg,, Bamberg
  - KPPK Studienzentrum Kroker-Schmidt, Bendorf
  - MECS Research GmbH, Berlin
  - Praxis Dr. Med Evelin Liefring, Berlin
  - Gemeinscharftspraxis Dres Jung - Deggingen, Deggingen
  - Medizentrum Essen Borbeck, Essen
  - Praxis Dr med Claus Keller, Frankfurt am Main
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Asklepios MVZ Bayern GmbH, Landsberg
  - Salvus-Klinische Studien GmbH, Leipzig
  - Zentrum fuer ambulante pneumologische Forschung Marburg GbR, Marburg
  - Studienzentrum Dr Med Schlenska, Peine
- Tuen Mun Hospital, Hong Kong, Hong Kong
- Israel (7):
  - Assuta Ashdod Medical Center, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Shamir Medical Center Assaf Harofeh, Beer Jacob
  - Tel Aviv Sourasky Medical Center PPDS, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center - PPDS, Tel Litwinsky
- Mexico (6):
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara, Jalisco
  - Centro de Investigacion Medico Biologico y Terapia Avanzada, S.C., Guadalajara, Jalisco
  - Unidad Medica de Occidente, Guadalajara, Jalisco
  - CICUM San Miguel, Guadalajara Centro, Jalisco
  - Unidad de Investigacion Clinica En Medicina (Udicem) S.C., Monterrey, Nuevo León
  - Centro de Investigacion y Atencion Integral Durango CIAID, Durango
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Isala Klinieken, Zwolle
- New Zealand (2):
  - Aotearoa Clinical Trials Trust, Auckland
  - Canterbury Respiratory Research Group, Christchurch
- Peru (4):
  - Clinica Providencia (Inverconsult Sociedad Anonima), Lima
  - Clinica Internacional, Lima
  - Clinica Ricardo Palma, Lima
  - Alfredo Berrocal Kasay Reuma Sociedad de Responsabilidad Limitada, Lima Cercado
- Poland (15):
  - Centrum Medyczne Bydgoszcz- PRATIA - PPDS, Bydgoszcz
  - Indywidualna Specjalistyczna Praktyka Lekarska lek., Kielce
  - Centrum Medyczne ALL-MED, Krakow
  - Diamond Clinic, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne ProMiMed sp z o.o. sp.k., Krakow
  - ETG Lodz, Lódz
  - ETG Lublin, Lublin
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól
  - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olec-Cudzik, Ostrowiec Swietokrzysk
  - Centrum Alergologii Teresa Hofman, Poznan
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów
  - ETG Siedlce, Siedlce
  - PULMAG Grzegorz Gasior Marzena Kociolek Spolka Cywilna, Sosnowiec
  - ETG Warszawa- PPDS, Warsaw
  - Dobrostan Gabinety Lekarskie, Wroclaw
- Romania (5):
  - Neomed Out-Patient Treatment and Diagnosis Medical Center SRL, Brasov
  - Dr. Victor Babes Foundation, Bucharest
  - Leon Daniello Pneumophthisiology Clinical Hospital, Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie Constanta, Constanța
  - Sf. Ioan cel Nou Emergency County Hospital, Suceava
- South Africa (6):
  - University of Cape Town Lung Institute, Cape Town
  - Clinical Trial Systems, City of Tshwane
  - St Augustines Hospital, Durban
  - Dr A.C Wilhase practice-Reimed, Ekurhuleni
  - Lakeview Hospital, Ekurhuleni
  - Langeberg Clinical Trials, Kraaifontein
- South Korea (4):
  - Catholic Univ. of Incheon St.Mary's Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Korea University Anam Hospital, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (9):
  - Hospital de Merida, Mérida, Badajoz
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - CHUS H Clinico U de Santiago, Santiago de Compostela, LA Coruna
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- Sweden (4):
  - Fysikalisk Medicin i Stockholm AB, Lidingö
  - ProbarE i Lund AB, Lund
  - PharmaSite, Malmo
  - ProbarE i Stockholm AB, Stockholm
- United Kingdom (5):
  - Queen Anne Street Medical Centre, London, London, City of
  - Bradford Royal Infirmary, Bradford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Ninewells Hospital, Dundee
  - Glenfield Hospital, Leicester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing